CLINICAL TRIAL: NCT04639362
Title: First Line Treatment With VeNEtoclaX and ibruTinib Induction Followed by Obinutuzumab intenSificaTion Exclusively in CLL/SLL Patients Not in Complete Remission and/or With Detectable Bone Marrow Minimal Residual Disease (NEXT STEP Trial)
Brief Title: CLL Induction Treatment With Venetoclax and Ibrutinib, Followed by Ibrutinib and Obinutuzumab in Patients With MRD.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Collaborators: Nordic Lymphoma Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HO158; 2019-002528-34 (EudraCT Number)
Record Dates: First submitted 2020-11-05; First posted 2020-11-20 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: CLL
MeSH Terms: interventions — ibrutinib; venetoclax; obinutuzumab; Observation

STUDY DESIGN:
Intervention Model Description: After 15 to 16 cycles of treatment the PI will assign patients to either observation (no further treatment) or intensification (treatment with ibrutinib and obinutuzumab), based on MRD results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensification (Experimental): Patients will receive 3 cycles lead-in with ibrutinib 420 mg/day. Here-after, patients will continue with 13 induction cycles (including one bridging cycle) combining ibrutinib 420 mg/day and venetoclax 400 mg/day (including a ramp up of 5 weeks). Patients who are not in CR or who have detectable MRD after 15 cycles (3 cycles lead-in and 12 cycles induction) will continue with 6 intensification cycles ibrutinib in combination with obinutuzumab day 1, 2, 8, 15 for the first cycle and with obinutuzumab day 1 for the following 5 cycles.
  Interventions: Drug: ibrutinib, venetoclax, obinutuzumab
- Observation (Experimental): Patients will receive 3 cycles lead-in with ibrutinib 420 mg/day. Here-after, patients will continue with 13 induction cycles (including one bridging cycle) combining ibrutinib 420 mg/day and venetoclax 400 mg/day (including a ramp up of 5 weeks). Patients who are in CR or have no detectable MRD will be observed.
  Interventions: Drug: ibrutinib, venetoclax

INTERVENTIONS:
Drug: ibrutinib, venetoclax, obinutuzumab — Patients will receive 3 cycles lead-in with ibrutinib 420 mg/day. Here-after, patients will continue with 13 induction cycles (including one bridging cycle) combining ibrutinib 420 mg/day and venetoclax 400 mg/day (including a ramp up of 5 weeks). Patients who are not in CR or who have detectable MRD after 15 cycles (3 cycles lead-in and 12 cycles induction) will continue with 6 intensification cycles ibrutinib in combination with obinutuzumab day 1, 2, 8, 15 for the first cycle and with obinutuzumab day 1 for the following 5 cycles.
  Other Names: Intensification
  Arms: Intensification
Drug: ibrutinib, venetoclax — Patients will receive 3 cycles lead-in with ibrutinib 420 mg/day. Here-after, patients will continue with 13 induction cycles (including one bridging cycle) combining ibrutinib 420 mg/day and venetoclax 400 mg/day (including a ramp up of 5 weeks). Patients who are in CR or have no detectable MRD will be observed.
  Other Names: Observation
  Arms: Observation

SUMMARY:
A recent study showed that 6 cycles of obinutuzumab when given after at least 1 year of ibrutinib did result in MRD conversion in a significant proportion of patients (50%). The precise influence, timing and interplay of venetoclax, ibrutinib and obinutuzumab on clearance of CLL cells in different compartments (PB, BM, LN), and achievement of uMRD and complete remission (CR) are not well known.

Therefore, the investigators set out a study to evaluate whether patients who are not in CR or who have detectable MRD after 12 months of combination treatment with ibrutinib and venetoclax (15 months total treatment including three months ibrutinib lead-in) could be converted into uMRD CR with an additional 6 cycles obinutuzumab in combination with ibrutinib.

DETAILED DESCRIPTION:
The BCL-2 antagonist venetoclax, specifically if combined with a CD20 antibody proved highly active in clearance of chronic lymphocytic leukemia (CLL) cells in peripheral blood (PB) and bone marrow (BM) but less so in lymph nodes (LN), probably due to the abundant expression of additional anti-apoptotic proteins within the LN compartment. The investigators hypothesize that due to the forced egress from the LN by ibrutinib, leukemic cells cannot escape from the apoptosis initiating effects of venetoclax, making combination of these drugs highly effective. Preliminary data from multiple ongoing trials on this combination are indeed promising, with not only superior rates of undetectable minimal residual disease (uMRD) than other ibrutinib combinations but perhaps more important, achievement of complete LN responses in the majority of patients. Yet, also with this combination, a significant subgroup of patients are expected to remain with detectable MRD. A recent study showed that 6 cycles of obinutuzumab when given after at least 1 year of ibrutinib did result in MRD conversion in a significant proportion of patients (50%). The precise influence, timing and interplay of venetoclax, ibrutinib and obinutuzumab on clearance of CLL cells in different compartments (PB, BM, LN), and achievement of uMRD and complete remission (CR) are not well known.

Therefore, the investigators set out a study to evaluate whether patients who are not in CR or who have detectable MRD after 12 months of combination treatment with ibrutinib and venetoclax (15 months total treatment including three months ibrutinib lead-in) could be converted into uMRD CR with an additional 6 cycles obinutuzumab in combination with ibrutinib. In addition to efficacy, as measured by undetectable MRD rate, emphasis of this trial will be on clearance of different compartments (PB, BM, LN) at different time points on protocol and in follow up. In addition, the toxicity profile is taken into consideration.

ELIGIBILITY:
Inclusion Criteria:

* Documented CLL or SLL requiring treatment according to IWCLL criteria33, including minimal required markers (CD5/CD19/CD23 triple positive with light chain restriction);
* WHO performance status 0-3 (appendix C), stage 3 only if attributable to CLL/SLL;
* No prior treatment for CLL/SLL;
* Age at least 18 years;
* Adequate BM function defined as:

  * Hb > 5 mmol/l or Hb > 8 g/dL
  * Absolute neutrophil count (ANC) ≥ 0.75 x 109/L or 750/μL
  * Platelet count ≥ 50 x 109/L or 50,000 /μL Unless directly attributable to CLL/SLL infiltration of the BM, proven by BM biopsy;
* Estimated Glomerular Filtration Rate (eGFR) (MDRD) or estimated creatinine clearance (CrCl) ≥ 30ml/min (Cockcroft-Gault appendix E); Please note: in case eGFR or CrCl is <50ml/min the patient needs to be considered high risk for TLS
* Adequate liver function as indicated:

  * Serum aspartate transaminase (ASAT) and alanine transaminase (ALAT) ≤ 3.0 x upper limit of normal (ULN)
  * Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of nonhepatic origin);
* Prothrombin time (PT)/International normal ratio (INR) <1.5 x ULN and activated partial thromboplastin time (aPTT) <1.5 x ULN;
* Negative serological testing for hepatitis B virus (Hepatitis B surface antigen (HBsAg) negative and hepatitis B core antibody (anti-HBc) negative) and hepatitis C virus (hepatitis C antibody). Subjects who are positive for hepatitis B core antibody, hepatitis B surface antigen, or hepatitis C antibody must have a negative PCR result before enrollment. Those who are PCR positive will be excluded;
* Ability and willingness to adhere to the study visit schedule and other protocol requirements;
* Patient is capable of giving informed consent;
* Written informed consent.

Exclusion Criteria:

* Transformation of CLL (Richter's transformation);
* Malignancies other than CLL/SLL currently requiring systemic therapy or not being treated in curative intention or showing signs of progression after curative treatment;
* Patient with CNS involvement
* Known allergy to xanthine oxidase inhibitors and/or rasburicase;
* Intolerance of exogenous protein administration;
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies. Known sensitivity or allergy to murine products;
* Active fungal, bacterial, and/or viral infection that requires systemic therapy; Please note: active controlled as well as chronic/recurrent infections are at risk of reactivation/infection during treatment (see section 9.2.3.1);
* Concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled: infection, auto-immune hemolysis, immune thrombocytopenia, diabetes, hypertension, hyperthyroidism or hypothyroidism etc.);
* Patients known to be HIV-positive;
* Patient requiring treatment with a strong cytochrome P450 (CYP) 3A inhibitor (see appendix K) or anticoagulant therapy with warfarin or phenprocoumon n or other vitamin K antagonists; Please note: Patients being treated with DOACs apixaban, edoxaban or rivaroxaban can be included, but must be properly informed about the potential risk of bleeding under treatment with ibrutinib. Treatment with dabigatran should be avoided, due to risk of toxicity based on P-gp substrate (see appendix K)
* History of stroke or intracranial hemorrhage within 6 months prior to registration;
* Severe cardiovascular disease (arrhythmias requiring chronic treatment, congestive heart failure or symptomatic ischemic heart disease) (CTCAE grade III-IV, see appendix D);
* Severe pulmonary dysfunction (CTCAE grade III-IV, see appendix D);
* Patient with Child Pugh C
* Severe neurological or psychiatric disease (CTCAE grade III-IV, see appendix D);
* Vaccination with live vaccines within 28 days prior to registration;
* Use of any other experimental drug or therapy within 28 days prior to registration
* Major surgery within 28 days prior to registration;
* Steroid therapy within 10 days prior to registration, with the exception of inhaled steroids for asthma, topical steroids, steroids up to 20 mg of dose equivalents of prednisolone daily to control autoimmune phenomenon's, or replacement/stress corticosteroids;
* Pregnant women and nursing mothers;
* Fertile men or women of childbearing potential unless: (1) surgically sterile or ≥ 2 years after the onset of menopause, and/or (2) willing to use a highly effective contraceptive method such as oral contraceptives, intrauterine device, sexual abstinence or barrier method of contraception in conjunction with spermicidal jelly during study treatment and in female patients for 3 months after end of induction treatment and 18 months after end of treatment with obinutuzumab and male patients for 6 months after end of treatment;
* Current participation in other clinical trial;
* Any psychological, familial, sociological and geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
BM uMRD CR 3 months after end of intensification with ibrutinib/obinutuzumab in patients who were not in CR or who had detectable MRD on combination ibrutinib and venetoclax. | 5 years
  Intensification arm

SECONDARY OUTCOMES:
BM uMRD CR 9 months after registration 2 in all subjects | 5 years
  Intensification arm
Best BM MRD level on protocol | 5 years
  Intensification arm
MRD level in BM and PB at different time points on protocol and in follow up | 5 years
  Intensification arm
Best response by IWCLL on protocol | 5 years
  Intensification arm
Response by IWCLL at different time points | 5 years
  Intensification arm
Response by Deauville criteria on PET scan at different time points | 5 years
  Intensification arm
Progression free survival (PFS), defined as time from registration 1 and from registration 2 to progression or death from any cause, whichever comes first | 5 years
  Intensification arm
Event free survival (EFS), defined as time from registration 1 and from registration 2 to start new CLL treatment, progression or death, whichever comes first | 5 years
  Intensification arm
Overall survival (OS), defined as time from registration 1 and from registration 2 to death from any cause | 5 years
  Intensification arm
Treatment free interval (TFI), defined as date of last protocol treatment to start date of first CLL treatment off protocol, or death from any cause whichever comes first | 5 years
  Intensification arm
Predictive value of prognostic markers at diagnosis on uMRD and ORR by IWCLL and Deauville criteria at end of ibrutinib/venetoclax and ibrutinib/obinutuzumab | 5 years
  Intensification arm
CTCAE grade ≥2 toxicities | 5 years
  Intensification arm
IWCLL hematological grade ≥2toxicities | 5 years
  Intensification arm

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Kater, PhD, Principal Investigator — Amsterdam UMC
Locations (27):
- Denmark (4):
  - DK-Aalborg-AALBORGUH, Aalborg
  - DK-Herlev-HERLEV, Herlev
  - DK-Odense-OUH, Odense
  - DK-Roskilde-ROSKILDE, Roskilde
- Netherlands (23):
  - NL-Almere-FLEVOZIEKENHUIS, Almere Stad
  - NL-Amersfoort-MEANDERMC, Amersfoort
  - NL-Amsterdam-AMC, Amsterdam
  - NL-Amsterdam-VUMC, Amsterdam
  - NL-Dordrecht-ASZ, Dordrecht
  - NL-Ede-ZGV, Ede
  - NL-Eindhoven-CATHARINA, Eindhoven
  - NL-Enschede-MST, Enschede
  - NL-Gouda-GROENEHART, Gouda
  - NL-Groningen-UMCG, Groningen
  - NL-Hilversum-TERGOOI, Hilversum
  - NL-Hoofddorp-SPAARNEGASTHUIS, Hoofddorp
  - NL-Roermond-LZR, Roermond
  - NL-Rotterdam-IKAZIA, Rotterdam
  - NL-Sittard-Geleen-ZUYDERLAND, Sittard
  - NL-Sneek-ANTONIUSSNEEK, Sneek
  - NL-Terneuzen-ZORGSAAM, Terneuzen
  - NL-Den Haag-HAGA, The Hague
  - NL-Den Haag-HMCWESTEINDE, The Hague
  - NL-Tilburg-ETZ, Tilburg
  - NL-Uden-BERNHOVEN, Uden
  - NL-Utrecht-UMCUTRECHT, Utrecht
  - NL-Zwolle-ISALA, Zwolle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kater AP, Kersting S, Dubois JM, van der Holt B, da Cunha-Bang C, Te Raa D, Idink C, de Boer F, Droogendijk J, de Heer K, van der Burg L, Nijziel MR, Tick L, Levenga H, Silbermann M, Ludwig I, Beeker A, Bellido M, Dobber JA, Evers LM, van der Kevie-Kersemaekers AM, Mellink C, Meulendijks I, Cunha S, Abrahamse-Testroote M, Zwezerijnen G, Zijlstra J, Niemann CU, Levin MD. Fixed-duration ibrutinib-venetoclax with MRD-guided ibrutinib-obinutuzumab intensification in first-line chronic lymphocytic leukaemia (HOVON 158/NEXT STEP): primary analysis of a multicentre, open-label, phase 2 trial. Lancet Haematol. 2025 Dec;12(12):e935-e945. doi: 10.1016/S2352-3026(25)00288-1. PMID 41338862
- See also: sponsor web site — http://www.hovon.nl